CLINICAL TRIAL: NCT06208878
Title: A Long-term Follow-up Study of Subjects With Malignancies Treated With CRISPR CAR T Cellular Therapies
Brief Title: A Long-term Follow-up Study of Subjects Who Received CRISPR CAR T Cellular Therapies
Status: Enrolling by invitation | Type: Observational
Sponsor: CRISPR Therapeutics AG (Industry)
Responsible Party: Sponsor
Organization: CRISPR Therapeutics (Industry)
Other Study IDs: CRSP-ONC-LTF
Record Dates: First submitted 2023-12-12; First posted 2024-01-17 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hematologic Malignancy; Solid Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non Interventional: All subjects with hematological and solid malignancies who are enrolled in a parent study and were exposed to allogeneic CRISPR CAR T cellular therapy will be asked to participate in this long-term follow-up (LTFU) study.
  Interventions: Other: Non Interventional

INTERVENTIONS:
Other: Non Interventional — Safety and Efficacy Assessment

SUMMARY:
This study will evaluate the long-term safety and efficacy of CRISPR CAR T cellular therapies

DETAILED DESCRIPTION:
All subjects with hematological and solid malignancies who are enrolled in a parent study and were exposed to allogeneic CRISPR CAR T cellular therapy will be asked to participate in this long-term follow-up (LTFU) study. Subjects who have completed the parent study for the protocol-defined duration, or who have discontinued the parent study early, or who are in secondary follow-up (follow up of subjects with progressive disease or who receive a subsequent line of anticancer therapy) in the parent study may enroll in this LTFU study. This will allow for collection of long-term efficacy data (as applicable) and safety data up to 15 years post-treatment with CRISPR CAR T cellular therapies.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with protocol-required study procedures and voluntarily sign and date a written informed consent document.
* Must have received CRISPR CAR T cellular therapy.

Exclusion Criteria:

* There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects with hematological and solid malignancies who are enrolled in a parent study and were exposed to allogeneic CRISPR CAR T cellular therapy will be asked to participate in this long-term follow-up (LTFU) study. Subjects who have completed the parent study for the protocol-defined duration, or who have discontinued the parent study early, or who are in secondary follow-up (follow up of subjects with progressive disease or who receive a subsequent line of anticancer therapy) in the parent study may enroll in this LTFU study. This will allow for collection of long-term efficacy data (as applicable) and safety data up to 15 years post-treatment with CRISPR CAR T cellular therapies.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2038-08 (Estimated); Study Completion 2038-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events, serious adverse events and adverse events of special interest related to CRISPR CAR T cellular therapy treatment. | 15 years
  The number and percentage of subjects with CRISPR CAR T cellular therapy related SAEs and AESIs will be summarized.

SECONDARY OUTCOMES:
The overall survival and duration of remission/response following CRISPR CAR T cellular therapy treatment | 15 years
  Overall survival will be calculated as the time between the initial dose of CRISPR CAR T cellular therapy in the parent study and death due to any cause. Duration of remission/response will be calculated as the time between the first objective response to first disease progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (17):
  - City of Hope, Duarte, California
  - Cedars Sinai, Los Angeles, California
  - Stanford, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Emory, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kansas, Westwood, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University Saint Louis, St Louis, Missouri
  - MSKCC, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Methodist Hospital-Sarah Cannon, San Antonio, Texas
  - University of Utah-Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - Sir Charles Gairdner, Nedlands
- Princess Margaret, Toronto, Ontario, Canada
- University Hospital Hamburg-Eppendorf, Hamburg, Germany